CLINICAL TRIAL: NCT04924075
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Belzutifan (MK-6482, Formerly PT2977) Monotherapy in Participants With Advanced Pheochromocytoma/Paraganglioma (PPGL), Pancreatic Neuroendocrine Tumor (pNET), Von Hippel-Lindau (VHL) Disease-Associated Tumors, Advanced Gastrointestinal Stromal Tumor (wt GIST), or Advanced Solid Tumors With HIF-2α Related Genetic Alterations
Brief Title: Belzutifan/MK-6482 for the Treatment of Advanced Pheochromocytoma/Paraganglioma (PPGL), Pancreatic Neuroendocrine Tumor (pNET), Von Hippel-Lindau (VHL) Disease-Associated Tumors, Advanced Gastrointestinal Stromal Tumor (wt GIST), or Solid Tumors With HIF-2α Related Genetic Alterations (MK-6482-015)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6482-015; MK-6482-015 (Other: MSD); PT2977 (Other: Former name); jRCT2011220024 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2023-504853-11-00 (Registry Identifier: EU CT); 2020-005028-13 (EudraCT Number)
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pheochromocytoma/Paraganglioma; Pancreatic Neuroendocrine Tumor; Von Hippel-Lindau Disease; Advanced Gastrointestinal Stromal Tumor; HIF-2α Mutated Cancers
Keywords: HIF-2α; Pheochromocytoma/paraganglioma; Pancreatic NET
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Adenoma, Islet Cell; von Hippel-Lindau Disease | interventions — belzutifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belzutifan (Experimental): Belzutifan, 120 mg, oral, once daily (QD) until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — Belzutifan, 120 mg, oral, once daily (QD) until progressive disease or discontinuation.
  Other Names: MK-6482; WELIREG™

SUMMARY:
This is a study to evaluate the efficacy and safety of belzutifan monotherapy in participants with advanced pheochromocytoma/paraganglioma (PPGL), pancreatic neuroendocrine tumor (pNET), von Hippel-Lindau (VHL) disease-associated tumors, advanced wt (wild-type) gastrointestinal stromal tumor (wt GIST), or advanced solid tumors with hypoxia inducible factor-2 alpha (HIF-2α) related genetic alterations. The primary objective of the study is to evaluate the objective response rate (ORR) of belzutifan per response evaluation criteria in solid tumors version 1.1 (RECIST 1.1) by blinded independent central review (BICR).

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Male and female participants at least 12 years of age (at least 18 years of age for Cohort B1)
* Diagnosis of one of the following: Advanced/metastatic pheochromocytoma/paraganglioma (PPGL), pancreatic neuroendocrine tumors (pNET), von Hippel-Lindau (VHL) disease associated localized tumors, or advanced wild-type gastrointestinal stromal tumor (wt GIST) or advanced solid tumors with Hypoxia Inducible Factor- 2 alpha subunit (HIF-2α) related genetic alterations
* Cohort BI: VHL Disease-associated tumors:

  * Have a diagnosis of VHL disease as determined by a germline test locally and/or clinical diagnosis
  * Must be ≥18 years of age
* Has a life expectancy of at least 3 months

The main exclusion criteria include but are not limited to the following:

* Unable to swallow orally administered medication or has a disorder that might affect the absorption of belzutifan
* History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* Any of the following: A pulse oximeter reading <92% at rest, or requires intermittent supplemental oxygen, or requires chronic supplemental oxygen
* Clinically significant cardiac disease, including unstable angina, acute myocardial infarction, or arterial bypass (CABG) or Percutaneous transluminal coronary angioplasty (PTCA) ≤6 months from study entry, or New York Heart Association Class III or IV congestive heart failure
* Received prior treatment (except somatostatin analogs) with chemotherapy, targeted therapy, biologics, or other investigational therapy within the past 4 weeks of first dose of study intervention

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2029-06-04 (Estimated); Study Completion 2029-06-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 5.5 years
  ORR is the percentage of participants with complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of the diameters of target lesions) until progressive disease (PD, at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progression) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Duration of Response (DOR) as Assessed by BICR | Up to approximately 5.5 years
  DOR is the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Time to Response (TTR) as Assessed by BICR | Up to approximately 5.5 years
  TTR is defined as the time from first dose of belzutifan to first documented evidence of CR or PR.
Disease Control Rate (DCR) as Assessed by BICR | Up to approximately 5.5 years
  Disease control is a confirmed CR, PR, or stable disease (SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study).
Progressive Free Survival (PFS) as Assessed by BICR | Up to approximately 5.5 years
  PFS is the time from first dose of belzutifan to the first documented PD or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 5.5 years
  OS is the time from first dose of belzutifan until death from any cause.
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 5.5 years
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Number of Participants Discontinuing Study Drug due to an AE | Up to approximately 5.5 years
  An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who discontinue study treatment due to an AE will be presented.
Time to Surgery (TTS) | Up to approximately 5.5 years
  TTS is defined as the time from the first dose of belzutifan to the first documented surgical intervention or tumor reduction procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (84):
- United States (14):
  - Cedars-Sinai Medical Center ( Site 0110), Los Angeles, California
  - Northwestern University - Robert H. Lurie Comprehensive Cancer Center ( Site 0130), Chicago, Illinois
  - Northwestern Medicine Cancer Center - Warrenville ( Site 0134), Warrenville, Illinois
  - University of Iowa ( Site 0104), Iowa City, Iowa
  - Johns Hopkins Hospital-Sidney Kimmel Comprehensive Cancer Center - Developmental Therapeutics ( Site 0108), Baltimore, Maryland
  - National Institutes of Health ( Site 0125), Bethesda, Maryland
  - Massachusetts General Hospital ( Site 0111), Boston, Massachusetts
  - University of Michigan ( Site 0126), Ann Arbor, Michigan
  - Washington University-Internal Medicine/Oncology ( Site 0124), St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai ( Site 0123), New York, New York
  - Penn Medicine: University of Pennsylvania Health System-Heme/Onc ( Site 0127), Philadelphia, Pennsylvania
  - SCRI Oncology Partners ( Site 7000), Nashville, Tennessee
  - Vanderbilt University Medical Center ( Site 0107), Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center ( Site 0112), Houston, Texas
- Australia (2):
  - Prince of Wales Hospital-Medical Oncology ( Site 1601), Randwick, New South Wales
  - The Royal Melbourne Hospital ( Site 1602), Parkville, Victoria
- Canada (2):
  - Arthur J.E. Child Comprehensive Cancer Centre ( Site 0203), Calgary, Alberta
  - Princess Margaret Cancer Centre ( Site 0202), Toronto, Ontario
- Chile (2):
  - FALP ( Site 2200), Santiago, Region M. de Santiago
  - Centro de Oncología de Precisión ( Site 2203), Santiago, Region M. de Santiago
- China (4):
  - Peking University First Hospital-Urology ( Site 1900), Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center ( Site 1905), Guangzhou, Guangdong
  - Renji Hospital Shanghai Jiao Tong University School of Medicine ( Site 1904), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University ( Site 1906), Chengdu, Sichuan
- Denmark (3):
  - Rigshospitalet ( Site 0304), Copenhagen, Capital Region
  - Rigshospitalet-Department of Endocrinology ( Site 0303), Copenhagen, Capital Region
  - Odense Universitetshospital ( Site 0302), Odense, Region Syddanmark
- France (6):
  - CHU Strasbourg-Hautepierre-Medecine Interne, Endocrinologie et Nutrition ( Site 0402), Strasbourg, Alsace
  - Hôpital Edouard Herriot-oncologie ( Site 0405), Lyon, Auvergne-Rhône-Alpes
  - Institut Paoli-Calmettes-Oncology ( Site 0406), Marseille, Bouches-du-Rhone
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre ( Site 0407), Le Kremlin-Bicêtre, Paris
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 0404), Paris
  - Gustave Roussy ( Site 0403), Villejuif, Île-de-France Region
- Germany (5):
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen-Department of Internal Medicine IV, Division ( Site 0501), München, Bavaria
  - Comprehensive Cancer Center Mainfranken-Div. of Endocrinology and Diabetes ( Site 0500), Würzburg, Bavaria
  - Universitaetsklinikum Freiburg ( Site 0504), Freiburg, Brandenburg
  - Universitaetsklinikum Duesseldorf-Gastroenterology, Hepatology and Infectiology ( Site 0505), Düsseldorf, North Rhine-Westphalia
  - Charité Universitaetsmedizin Berlin - Campus Mitte-Department of Endocrinology and Metabolism ( Site 0503), Berlin
- Semmelweis University-Belgyógyászati és Onkológiai Klinika Hematológia Osztály ( Site 0600), Budapest, Hungary
- Israel (2):
  - Sheba Medical Center-Institute of Endocrinology, Diabetes and Metabolism ( Site 1400), Ramat Gan
  - Sourasky Medical Center ( Site 1401), Tel Aviv
- Italy (8):
  - University of Naples Federico II-Dipartimento di Medicina Clinica e Chirurgia ( Site 0704), Naples, Campania
  - Fondazione IRCCS Istituto Nazionale dei Tumori-S.C. Oncologia Medica 2- Sarcomi ( Site 0709), Milan, Lombardy
  - Azienda Ospedaliero Universitaria Senese-U.O.C. Immunoterapia Oncologica ( Site 0706), Siena, Tuscany
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 0708), Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia-Oncology ( Site 0701), Brescia
  - Ospedale San Raffaele-Oncologia Medica ( Site 0705), Milan
  - Istituto Europeo di Oncologia IRCCS-Divisione di Oncologia Medica Gastrointestinale e Tumori Neuroe ( Site 0700), Milan
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma ( Site 0703), Verona
- Japan (6):
  - Hokkaido University Hospital ( Site 1800), Sapporo, Hokkaido
  - Yokohama City University Hospital ( Site 1804), Yokohama, Kanagawa
  - Kochi Medical School Hospital ( Site 1807), Nankoku, Kochi
  - National Cancer Center Hospital ( Site 1802), Chuo-ku, Tokyo
  - Kyoto University Hospital ( Site 1806), Kyoto
  - Tokyo Women's Medical University Adachi Medical Center ( Site 1803), Tokyo
- Universitair Medisch Centrum Utrecht ( Site 1530), Utrecht, Netherlands
- Oslo Universitetssykehus Radiumhospitalet ( Site 2400), Oslo, Norway
- Portugal (2):
  - START Lisbon - Hospital de Santa Maria ( Site 2601), Lisbon, Lisbon District
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil E.P.E. ( Site 2600), Porto
- Russia (5):
  - GBUZ Republican Clinical Oncological Dispensary ( Site 0804), Ufa, Baskortostan, Respublika
  - Saint Petersburg State University-Clinic of advanced medical technologies n. a. Nicolay I. Pirogov ( Site 0805), Saint Petersburg, Leningradskaya Oblast'
  - Saint-Petersburg City Clinical Oncology Dispensary-Department of chemotherapy ( Site 0803), Saint Petersburg, Leningradskaya Oblast'
  - Fed State Budgetary Inst N.N. Blokhin Med Center of Oncology MHRF ( Site 0801), Moscow, Moscow
  - Endocrinology Research Center of Rosmedtechnologies-Surgery ( Site 0809), Moscow, Moscow
- National Cancer Centre Singapore ( Site 1700), Singapore, Central Singapore, Singapore
- South Korea (2):
  - Seoul National University Hospital ( Site 2001), Jongno-gu, Seoul
  - Asan Medical Center ( Site 2000), Songpa-gu, Seoul
- Spain (4):
  - MD Anderson Cancer Center-Oncology ( Site 1102), Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre-Medical Oncology ( Site 1103), Madrid, Madrid, Comunidad de
  - Hospital Universitario Central de Asturias-Medical Oncology ( Site 1101), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron ( Site 1100), Barcelona
- Sweden (4):
  - Skanes University Hospital Lund ( Site 1200), Lund, Skåne County
  - Karolinska Universitetssjukhuset Solna ( Site 1202), Stockholm, Stockholm County
  - Akademiska sjukhuset-Blod- och tumörsjukdomar ( Site 1201), Uppsala, Uppsala County
  - Sahlgrenska Universitetssjukhuset-Department of Oncology CTU Clinical Trial Unit ( Site 1204), Gothenburg, Västra Götaland County
- Turkey (Türkiye) (5):
  - Baskent University Adana Training Hospital ( Site 0906), Yüreğir, Adana
  - Ege University Medicine of Faculty ( Site 0900), Bornova, İzmir
  - Hacettepe Universitesi-oncology hospital ( Site 0901), Ankara
  - Ankara Bilkent Şehir Hastanesi. ( Site 0904), Ankara
  - Istanbul Universitesi Cerrahpasa-Medical Oncology ( Site 0902), Istanbul
- United Kingdom (4):
  - Addenbrooke's Hospital ( Site 1309), Cambridge, Cambridgeshire
  - Royal Free Hospital ( Site 1302), London, England
  - The Beatson West of Scotland Cancer Centre ( Site 1308), Glasgow, Glasgow City
  - Hammersmith Hospital-Medical Oncology ( Site 1304), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Jimenez C, Andreassen M, Durand A, Moog S, Hendifar A, Welin S, Spada F, Sharma R, Wolin E, Ruether J, Garcia-Carbonero R, Fassnacht M, Capdevila J, Del Rivero J, Iliopoulos O, Huillard O, Jang R, Mai K, Artamonova E, Hallqvist A, Else T, Odeleye-Ajakaye A, Gozman A, Naik GS, Berruti A; LITESPARK-015 Investigators. Belzutifan for Advanced Pheochromocytoma or Paraganglioma. N Engl J Med. 2025 Nov 20;393(20):2012-2022. doi: 10.1056/NEJMoa2504964. Epub 2025 Oct 18. PMID 41124218
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26327&tenant=MT_MSD_9011